

## NCT# 02919111

# Gallium-68 PSMA-11 PET in intermediate to high-risk preprostatectomy patients

Protocol Number: CC #16559 Study Drug: Gallium-68 PSMA-11

Version Number: Version 1.1 Version Date: 6/8/2018

**IND Number: 127621** 

#### Principal Investigator (Sponsor-Investigator)

Thomas Hope, MD University of California San Francisco

#### **Co-Investigators**

Dr. Rahul Aggarwal, MD

Dr. Peter Carroll, MD

Dr. Matthew Cooperberg, MD

Dr. Michael Evans, PhD

Dr. Felix Feng, MD

Dr. Larry Fong, MD

Dr. Terence Friedlander, MD

Dr. Kirsten Greene, MD

Dr. John Kurhanewicz, PhD

Dr. Amy Lin, MD

Dr. Hao Nguyen, MD

Dr. Mack Roach, MD

Dr. Eric Small, MD

Dr. Li Zhang, PhD (Statistician)

#### **Clinical Research Coordinator**



#### **Proprietary and Confidential**



## **Protocol Signature Page**

Protocol No.: 16559 Version Date: 6/8/2018

- 1. I agree to follow this protocol version as approved by the UCSF Protocol Review Committee (PRC), Committee on Human Research (CHR), and Data Safety Monitoring Committee (DSMC).
- 2. I will conduct the study in accordance with applicable CHR requirements, Federal regulations, and state and local laws to maintain the protection of the rights and welfare of study participants.
- 3. I certify that I, and the study staff, have received the requisite training to conduct this research protocol.
- 4. I have read and understand the information in the Investigators' Brochure (or Manufacturer's Brochure) regarding the risks and potential benefits. I agree to conduct the protocol in accordance with Good Clinical Practices (ICH-GCP), the applicable ethical principles, the Statement of Investigator (Form FDA 1572), and with local regulatory requirements. In accordance with the FDA Modernization Act, I will ensure the registration of the trial on the www.clinicaltrials.gov website.
- 5. I agree to maintain adequate and accurate records in accordance with CHR policies, Federal, state and local laws and regulations.

| Thomas A. Hope | |
|----------------|-------------|
| Printed Name | <del></del> |
| Signature | Date |

**UCSF Principal Investigator / Study Chair** 

## **Abstract**

| Title | Gallium-68 PSMA-11 PET in patients with biochemical recurrence |
|---|---|
| Patient population | <ul> <li>Intermediate to high-risk disease (as determined by elevated PSA [PSA&gt;10], T-stage [T2b or greater], Gleason score [Gleason score &gt; 6] or other risk factors).</li> </ul> |
| Rationale for<br>Study | Gallium-68 PSMA-11 has been shown to have a higher sensitivity for the detection of metastatic prostate cancer compared to choline based imaging. |
| Primary<br>Objective | Sensitivity, specificity, positive and negative predictive value of PSMA PET for the detection of regional nodal metastases compared to pathology at radical prostatectomy on a per patient basis using nodal regional correlation. |
| Secondary<br>Objectives | <ul> <li>Sensitivity, specificity, positive and negative predictive value of PSMA PET for the detection of extra-pelvic nodal metastases, visceral metastases and osseous metastases compared to biopsy and imaging follow-up.</li> <li>Safety.</li> </ul> |
| Exploratory<br>Endpoints | Sensitivity, specificity, negative and positive predictive value for detection of regional nodal metastases in comparison to cross sectional imaging performed contemporaneously with the PSMA-11 PET. |
| | One year PSA progression free survival, comparing patients with and without pelvic nodal metastases. |
| | Correlation between SUV <sub>max</sub> from PSMA-11 PET and short axis diameter of nodal disease on cross sectional imaging correlate to presence of true pathology. |
| | Incidence of osseous and distant metastatic lesions. |
| Study Design | This is a phase 2/3 multi-center open label study. |
| Number of | Total population of patients will be 300 patients across all institutions. |
| patients | 300 patients imaged at UCSF. |
| Duration of<br>Therapy | The study will involve a single imaging study. |
| Duration of Follow up | The patients will be followed-up by phone one to three days after the study completion. |
| Duration of study | The study will reach completion three years from the time the study opens to accrual. |

| Study Drugs | callium-68 labeled PSMA-11 (or HBED-CC PSMA, DFKZ-11 or the eidelberg compound) |
|---|---|
| Safety<br>Assessments | Patient vital signs will be taken immediately before and after the administration of the radiopharmaceutical. The patients will also be asked to report adverse events. |

#### List of Abbreviations

AE adverse event

CHR Committee on Human Research (UCSF IRB)

CRC Clinical Research Coordinator

CRF case report form

CT computerized tomography

CTCEA Common Terminology Criteria for Adverse Events

DSMC Data and Safety Monitoring Committee

DSMP Data and Safety Monitoring Plan

ECOG Eastern Cooperative Oncology Group

FDA Food and Drug Administration

Ga-68 Gallium 68

HDFCCC Helen Diller Family Comprehensive Cancer Center

ICH International Conference on Harmonization

IND investigational new drug application

IRB Institutional Review Board

IV intravenous

MRI magnetic resonance imaging NCI National Cancer Institute

PET Positron Emission Tomography

PK pharmacokinetics

PRC Protocol Review Committee (UCSF)

PSA Prostate specific antigen

PSMA Prostate specific membrane antigen

SD standard deviation

## **Table of Contents**

| Pro | otocol Signature Page | 0 |
|---|---|---|
| Abs | stract 1 | |
| List | t of Abbreviations | 3 |
| | ble of Contents | |
| 1 | Introduction | |
| ' | | |
| | 1.1 Overview | |
| | 1.3 Patient Population | |
| 2 | Objectives of the Study | |
| | 2.1 Primary | |
| | 2.2 Secondary | |
| | 2.3 Exploratory | |
| | 2.4 Endpoints | |
| | 2.4.1 Primary Endpoints | |
| | 2.4.2 Secondary endpoints | 8 |
| | 2.4.3 Exploratory Endpoints | |
| 3 | Study Design | 8 |
| | 3.1 Characteristics | 8 |
| | 3.2 Number of Subjects | |
| | 3.3 Eligibility Criteria | |
| | 3.3.1 Inclusion Criteria | |
| | 3.3.2 Exclusion Criteria | |
| | 3.4 Duration of Follow Up | |
| | 3.5 Study Timeline | |
| | 3.5.1 Primary Completion | |
| 4 | Study Drugs | |
| • | • • | |
| | 4.1 Description, Supply and Storage of Investigational Drugs 4.1.1 Investigational Drug #1 | |
| 5 | Treatment Plan | |
| - | 5.1 Dosage and Administration | 9 |
| | 5.1.1 Other Modality(ies) or Procedures | ••••••••••• |
| | 5.2 Monitoring and Toxicity Management | |
| 6 | Study Procedures and Observations (Appendix 2 and 3) | |
| | 6.1 Schedule of Procedures and Observations | |
| | 6.1.2 Treatment Period | |
| | 6.1.3 Site level image interpretation | |
| | 6.1.4 Clinical follow-up | |
| | 6.1.5 Post-treatment Follow Up Visits | |
| | 6.2 Prohibited Medications | |
| 7 | Reporting and Documentation of Results | 12 |
| | 7.1 Evaluation of Efficacy (or Activity) | 12 |
| | 7.2 Evaluation of Safety | 12 |
| | 7.3 Definitions of Adverse Events | 12 |

## **Table of Contents**

| | 7.3. | .1 Adverse Event | 12 |
|------|-----------------|-----------------------------------------------|----|
| | 7.3. | | |
| | 7.4 | Recording of an Adverse Event | 13 |
| | 7.5 | Follow-up of Adverse Events | |
| | 7.6 | Expedited Reporting | 14 |
| 8 | Statistic | al Considerations and Evaluation of Results | 15 |
| | 8.1 | Study Endpoints | 15 |
| | 8.1. | * * | |
| | 8.2 | Determination of Sample Size and Accrual Rate | 15 |
| | 8.2. | .1 Sample Size and Power Estimate | 15 |
| | 8.2. | .2 Accrual estimates | 16 |
| | 8.3 | Analyses Plans | 16 |
| | 8.3. | .1 Analysis Population | 16 |
| | 8.3. | J J I | |
| | 8.3. | | |
| _ | 8.3. | | 20 |
| 9 | Study M | lanagement | 21 |
| | 9.1 | Pre-study Documentation | 21 |
| | 9.2 | Institutional Review Board Approval | 21 |
| | 9.3 | Informed Consent | |
| | 9.4 | Changes in the Protocol | |
| 10 | Protection | on of Human Subjects | 21 |
| Ref | 10.1<br>erences | Protection of Privacy23 | 21 |
| App | endices | 25 | |
| App | endix 1 | Performance Status Criteria | 25 |
| App | endix 2 | Schedule of procedures | 26 |
| | | ow chart) | |
| List | of Tables | | |
| Tal | ole 1.1 | Schedule of Study Procedures and Assessments | 26 |

## 1 Introduction

#### 1.1 Overview

Imaging and staging of prostate cancer is critical for surgical and treatment planning. We aim to image patients with suspected metastatic prostate cancer using Gallium-68 labeled HBED-CC PSMA (68Ga-PSMA-11) in order to demonstrate its utility. We plan to utilize this data to obtain further approvals of the 68Ga-PSMA-11compound, so that this agent will become available for clinical imaging in prostate cancer patients.

This compound has been shown to be superior to choline based PET agents for the staging of prostate cancer, both Carbon-11 and Fluorine-18 compounds. But this compound was not patented and therefore no company or private entity will make the investment required to bring <sup>68</sup>Ga-PSMA-11 to market. In the vacuum of availability, academic groups must take the lead in order to collect the necessary data for future FDA approval.

The rate of prostatectomy is increasing in high-risk prostate cancer patients (1), which means that there is an increasing unmeet need to detect regional and distant metastases prior to surgery. There have been two published studies looking in intermediate to high-risk patients using <sup>68</sup>Ga-PSMA-11 PET prior to prostatectomy, demonstrating a per patient sensitivity for nodal metastases of 64-66% (2,3), much improved compared to conventional imaging modalities. We aim to study the ability of <sup>68</sup>Ga-PSMA-11 to detect pelvic nodal disease in intermediate and high-risk preprostatectomy patients.

## 1.2 Background

Prostate cancer is the most commonly diagnosed cancer and second leading cause of cancer death in American men (1). Existing conventional imaging (CT, MRI and bone scans) has a low sensitivity in detecting local recurrence or metastatic disease (2). The one exception being NaF PET/CT for the detection of osseous metastasis. Due to this limitation, numerous approaches to stage patients have been evaluated.

Choline imaging has been frequently used, as prostate cancer exhibits increase choline uptake that has been associated with the presence of choline kinase (3). Choline uptake is increased in comparison to FDG in both androgen dependent and independent prostate cancer patients (4). Choline has also been shown to be sensitive for the detection of recurrent tumor in patients with PSA (prostate specific antigen) values of less than 1.0 ng/ml (5). There are two forms of choline that are used in imaging prostate cancer, C-11 and F-18 choline. C-11 choline has a short half-life of 20 minutes, which limits its detection for metastatic disease but results in improved local detection due to decreased urinary activity at the time of imaging. F-18 choline has significant urinary excretion that limits evaluation of the prostate but, but has been shown to have better detection rates for distant metastatic disease (6). C-11 choline has limited sensitivity for osseous metastasis, possibly due to the decreased uptake time (7). Additionally, the sensitivity of C-11 choline is limited in patients with PSA values < 1.0 ng/ml (8-10). Although choline PET may be limited in sensitivity, it clearly delineates more lesions than cross section imaging or bone scan in patients with known disease (11). In 2012, the Mayo Clinic obtained NDA (new drug application) approval from the FDA for the use of C-11 choline.

A separate approach is to image the prostate specific membrane antigen (PSMA). PSMA is expressed on the majority of prostate cancer cells, and so would be an ideal cell membrane protein to image. The initial imaging approach to PSMA imaging target the intracellular domain using Indium-111-capromab (Prostascint), a murine monoclonal antibody (12,13). Although there was early promise for the detection of nodal metastasis (14), the agent was never able to adequately visualize osseous metastasis (15). Although combination with SPECT/CT does improve lesion detection (16). One main limitation to In-111-capromab is that it takes a prolonged time to localize to the target tissue, which likely relates to both the size of the monoclonal antibody and the fact that agent targets the intracellular domain of the PSMA

protein. Additionally, Prostascint also recognizes an intracellular epitope so the antibody must cross the membrane to be effective. This likely only occurs in permeable dead or dying tumor cells.

Because of the limitations of In-111 capromab, there has been continued effort to develop agents that target the extracellular domain of the PSMA protein. The Ga-68 labeled PSMA-11 compound has become of particular interest because in the last year there have been two important articles. The first demonstrates that PSMA-11 has a higher sensitivity for the detection of disease than F-18 choline in a head-to-head intra-patient comparison that included 37 patients (17). The second paper looked at the sensitivity of PSMA-11 in the detection of metastatic lesions in patients with recurrent prostate cancer (18). Their results demonstrated a detection rate of 50% for patients with a PSA less than 1 ng/ml, and detection rate above 85% for patients with a PSA greater than 2 ng/ml. These detection rates are significantly higher than that reported by groups using choline (5).

Because of the improved resolution and image quality with PET, ability to quantitate uptake, increased sensitivity compared to choline, we intend to evaluate the utility of <sup>68</sup>Ga-PSMA-11 for the imaging of prostate cancer. We expect that the data from this study will support applications for clinical approval of this imaging agent, leading to wider availability within the United States.

## 1.3 Patient Population

Patients with intermediate to high-risk prostate cancer planning to undergo prostatectomy.

## 2 Objectives of the Study

## 2.1 Primary

Sensitivity, specificity, positive and negative predictive value of PSMA PET for the
detection of regional nodal metastases compared to pathology at radical prostatectomy
on a per patient basis using nodal regional correlation.

## 2.2 Secondary

- Sensitivity, specificity, positive and negative predictive value of PSMA PET for the
  detection of extra-pelvic nodal metastases, visceral metastases and osseous
  metastases compared to biopsy and imaging follow-up.
- Safety, as characterized by CTCAE 4.03.

#### 2.3 Exploratory

- Sensitivity, specificity, negative and positive predictive value for detection of regional nodal metastases in comparison to cross sectional imaging performed contemporaneously with the PSMA-11 PET.
- One year PSA progression free survival, comparing patients with and without pelvic nodal metastases.
- Correlation between SUV<sub>max</sub> from PSMA-11 PET and short axis diameter of nodal disease on cross sectional imaging correlate to presence of true pathology.
- Incidence of osseous and distant metastatic lesions.

#### 2.4 Endpoints

## 2.4.1 Primary Endpoints

- PSMA PET results for regional nodal disease.
  - Nodal histology results from prostatectomy.

## 2.4.2 Secondary endpoints

- PSMA PET results for extra-pelvic disease.
- Biopsy results and imaging follow-up results

## 2.4.3 Exploratory Endpoints

- Time to PSA progression
- SUV<sub>max</sub> of lesions.
- Presence of osseous and distant metastasis.
- Safety: blood pressure, heart rate, self reported adverse events

## 3 Study Design

#### 3.1 Characteristics

This is a prospective, multi-center, open-label study in patients with prostate cancer. Eligible participants will undergo baseline assessments at enrollment. Study participants will receive a one-time administration of Ga-68 PSMA-11 and undergo a PET/CT or PET/MRI imaging study.

#### 3.2 Number of Subjects

A total of 300 patients will be enrolled across all sites. 300 patients will be imaged at UCSF.

## 3.3 Eligibility Criteria

Patients must have baseline evaluations performed prior to the administration of the radiopharmaceutical and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent must be obtained from the patient prior to enrollment. The following criteria apply to all patients enrolled onto the study:

## 3.3.1 Inclusion Criteria

- 1. Biopsy proven prostate adenocarcinoma.
- 2. Planned prostatectomy with lymph node dissection.
- 3. Intermediate to high-risk disease (as determined by elevated PSA [PSA>10], T-stage [T2b or greater], Gleason score [Gleason score > 6] or other risk factors).
- 4. Karnofsky performance status of ≥50 (or ECOG/WHO equivalent).
- 5. Age > 18.
- 6. Ability to understand a written informed consent document, and the willingness to sign it.

#### 3.3.2 Exclusion Criteria

- 1. Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam.
- 2. Neoadjuvant chemotherapy or radiation therapy prior to prostatectomy.
  - a. Including focal ablation techniques (HiFu).

3. Androgen deprivation therapy or other neoadjuvant treatments prior to PET imaging and surgery.

4. Contraindication to furosemide administration including prior allergy or adverse reaction to furosemide or sulfa drugs. (Note: This exclusion criteria can be removed if Furosemide is omitted as part of the PET imaging protocol if a second-generation scatter correction is available for the used PET device).

## 3.4 Duration of Follow Up

Patients will be followed for one to three day after the administration of the radiopharmaceutical.

## 3.5 Study Timeline

## 3.5.1 Primary Completion

The study will reach primary completion 36 months from the time the study opens to accrual.

## 3.5.2 Study Completion

The study will reach study completion 48 months from the time the study opens to accrual.

## 4 Study Drugs

#### 4.1 Description, Supply and Storage of Investigational Drugs

## 4.1.1 Investigational Drug #1

Ga-68 labeled PSMA-11 (or PSMA-HBED-CC) is a radiopharmaceutical that will be produced under cGMP.

#### 5 Treatment Plan

## 5.1 Dosage and Administration

The imaging agent (Ga-68 PSMA-11 or PSMA-HBED-CC) will be administered on an outpatient basis. It will be administered a single time intravenously prior to the PET/CT imaging. The injected dose will be 3 to 7 mCi of <sup>68</sup>Ga-PSMA-11.

## 5.1.1 Other Modality(ies) or Procedures

#### **5.1.1.1 PET imaging**

- a) <sup>68</sup>Ga-PSMA-11 PET preparation and injection: The injected dose will be 111-259 MBq (3-7 mCi) of <sup>68</sup>Ga-PSMA-11 PET. A dose of 20 mg of Furosemide is recommended to be injected together with, shortly before or after administration of the radiotracer in order to minimize PET scatter artifacts from excreted radiotracer accumulation in the kidney and urinary bladder that can occur with PSMA-11. Oral hydration and voiding is recommended prior to the start of the scan. Furosemide should not be administered in patients with medical contraindications to furosemide administration including allergies and adverse reactions including sulfa allergies. (Note: Application of Furosemide can be omitted as part of the PET imaging protocol if a second-generation scatter correction algorithm is available for the PET scanner used in this protocol). PET imaging will begin 50-100 minutes after injection.
- b) PET protocol: Scan coverage will extend from mid thigh to the base of the skull, starting from the mid-thighs to prevent urinary bladder radiotracer accumulation at the start of PET imaging. Bed position scan time will be dependent on each sites scanner capabilities. At a minimum, 3 minutes per bed position will be used. In certain

circumstances, coverage may be extended to the toes. Contrast may be administered if requested by the referring clinician and is decided site dependent.

- i) If the patient has not had a diagnostic CT or MRI within one month of the <sup>68</sup>Ga-PSMA-11 PET, then <sup>68</sup>Ga-PSMA-11 PET study will be performed with a diagnostic CT or MRI.
- c) Safety monitoring: Vital signs will be assessed immediately before and after injection of <sup>68</sup>Ga-PSMA-11 (HR and supine BP). Patients will be monitored for adverse events during injection and for two hours after radiotracer administration. Additionally, patient's vitals (HR and supine BP) will be checked at the completion of the imaging study prior to leaving the imaging center.
- d) Patient follow-up: Patients will be contacted by phone one to three working days after <sup>68</sup>Ga-PSMA-11 PET to assess for the development of delayed adverse events. Patients will be seen in the clinic if there are any concerning study related adverse events requiring further evaluation.

## 5.2 Monitoring and Toxicity Management

Each patient receiving Ga-68 PSMA-11 will be evaluable for safety. The safety parameters include physical findings and spontaneous reports of adverse events reported to the investigator by patients.

## 6 Study Procedures and Observations (Appendix 2 and 3)

#### 6.1 Schedule of Procedures and Observations

Screening assessments must be performed within 30 days prior to the first dose of investigational product. Any results falling outside of the reference ranges may be repeated at the discretion of the investigator. Treatment or visit delays for public holidays or weather conditions do not constitute a protocol violation.

A written, signed, informed consent form (ICF) and a Health Insurance Portability and Accountability Act (HIPAA) authorization must be obtained before any study-specific assessments are initiated. A copy of the signed ICF will be given to the subject and a copy will be filed in the medical record. The original will be kept on file with the study records.

### **6.1.1.1 Screening Assessments**

The Screening procedures and assessments must be completed within 30 days of the day 1 Visit.

- Laboratory values: all patients must have a recent PSA (preferably within 30 days prior to the <sup>68</sup>Ga-PSMA-11 PET)
- Pathology: all patients must have histopathology/biopsy of the prostate with a documented Gleason score
- Performance status: all patients must have their Karnofsky performance status (or ECOG/WHO equivalent) evaluated (Appendix 1).

#### 6.1.2 Treatment Period

## 6.1.2.1 Study Procedures, Imaging Day 1

- Vital signs
- Evaluation of adverse events

## 6.1.3 Site level image interpretation

PET images will initially be interpreted by a board certified nuclear medicine physician or a board certified radiologist experienced in reading PET at the time of the imaging study at the institution that the study is being performed. These interpretations will not be used for final evaluation.

## 6.1.4 Clinical follow-up

- a) Prostatectomy: patients without evidence of PSMA-11 PET positive nodal or metastatic disease noted on imaging will undergo radical prostatectomy. If a PSMA-11 PET positive regional pelvic node is noted, the urologist will be informed of the location of the suspicious node and the patient will undergo prostatectomy with nodal dissection.
  - i) Patients with nodes seen on PSMA-11 PET without positive nodes on pathology, will be rescanned with CT or MRI to determine if the suspicious node was thought to be removed. A PSMA-11 PET may be repeated as well at the discretion of the treating physician.
- b) If sites of PSMA PET positive osseous or distant metastatic lesions are noted, the urologist will be informed, and further evaluation including further imaging (bone scan, NaF PET, CT or MRI cross section imaging) or targeted biopsy will be performed in order to restage the patient prior to the decision regarding whether or not a prostatectomy will be performed as per the responsible surgeon and standard of clinical care.

## 6.1.5 Post-treatment Follow Up Visits

Patients will be followed for one to three days after enrollment, by phone. The following procedure will be performed at 1-3 days:

Evaluation of adverse events

#### 6.2 Prohibited Medications

There are no prohibited medications.

## 7 Reporting and Documentation of Results

## 7.1 Evaluation of Efficacy (or Activity)

#### 7.1.1.1 Definitions

#### **Evaluable for toxicity**

All patients will be evaluable for toxicity from the time of Ga-68 PSMA-11.

## 7.2 Evaluation of Safety

Analyses will be performed for all patients receiving Ga-68 PSMA-11. The study will use the CTCAE v4.0 for reporting of adverse events.

## 7.3 Definitions of Adverse Events

#### 7.3.1 Adverse Event

An adverse event (also known as an adverse experience) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. More specifically, an adverse event (can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. An adverse event can arise from any use of the drug (e.g., off-label use, use in combination with another drug) and from any route of administration, formulation, or dose, including an overdose.

#### 7.3.2 Adverse reaction

An adverse reaction is defined as any adverse event caused by the use of a drug. Adverse reactions are a subset of all suspected adverse reactions for which there is reason to conclude that the drug caused the event.

#### 7.3.2.1 Suspected

A suspected adverse reaction is defined as any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of IND safety reporting, "reasonable possibility" indicates that there is evidence to suggest a causal relationship between the drug and the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 7.3.2.2 Unexpected

An adverse event or suspected adverse reaction is considered *unexpected* if it is not listed in the investigator brochure or package insert(s), or is not listed at the specificity or severity that has been observed, or, if an investigator brochure is not required or available, is not consistent with the risk information described in the general investigational plan or elsewhere in the current application.

"Unexpected," as used in this definition, also refers to adverse events or suspected adverse reactions that are mentioned in the investigator brochure as occurring with a class of drugs or

as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation.

Adverse events that would be anticipated to occur as part of the disease process are considered *unexpected* for the purposes of reporting because they would not be listed in the investigator brochure. For example, a certain number of non-acute deaths in a cancer trial would be anticipated as an outcome of the underlying disease, but such deaths would generally not be listed as a suspected adverse reaction in the investigator brochure.

#### 7.3.2.3 Serious

An adverse event or suspected adverse reaction is considered *serious* if, in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Death
- Life-threatening adverse event
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life function
- Congenital anomaly/birth defect

Important medical events that may not result in death, are life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

#### 7.3.2.4 Life-threatening

An adverse event or suspected adverse reaction is considered *life-threatening* if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

## 7.4 Recording of an Adverse Event

All grade 3 and above adverse events will be recorded using the NCI CTCAE v4.0. The Investigator will assign attribution of the possible association of the event with use of the investigational drug.

| Relationship | Attribution | Description |
|---|---|---|
| Unrelated to investigational | Unrelated | The AE <i>is clearly NOT related</i> to the intervention |
| drug/intervention | Unlikely | The AE <i>is doubtfully related</i> to the intervention |
| Deleted to investigation of | Possible | The AE may be related to the intervention |
| Related to investigational drug/intervention | Probable | The AE is likely related to the intervention |
| drug/intervention | Definite | The AE is clearly related to the intervention |

Signs or symptoms reported as adverse events will be graded and recorded by the Investigator according to the CTCAE. When specific adverse events are not listed in the CTCAE they will be graded by the Investigator as *none*, *mild*, *moderate* or *severe* according to the following grades and definitions:

- Grade 0 No AE (or within normal limits)
- Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
- Grade 2 Moderate; minimal, local, or noninvasive intervention (e.g., packing, cautery) indicated; limiting age-appropriate instrumental activities of daily living (ADL)
- Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL
- Grade 4: Life-threatening consequences; urgent intervention indicated
- Grade 5: Death related to AE

## 7.5 Follow-up of Adverse Events

All adverse events will be followed with appropriate medical management until resolved. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event. For selected adverse events for which administration of the investigational drug was stopped, a re-challenge of the subject with the investigational drug may be conducted if considered both safe and ethical by the Investigator.

## 7.6 Expedited Reporting

#### Reporting to the Data and Safety Monitoring Committee

If a death occurs during the treatment phase of the study or within 30 days after the last administration of the study drug(s) and it is determined to be related either to the study drug(s) or to a study procedure, the Investigator or his/her designee must notify the DSMC Chair (or qualified alternate) within 1 business day of knowledge of the event. The contact may be by phone or e-mail.

#### Reporting to UCSF Committee on Human Research (Institutional Review Board)

The Principal Investigator must report events meeting the UCSF CHR definition of "Unanticipated Problem" (UP) and the San Francisco VA Medical Center within 5 business days of his/her awareness of the event.

#### **Expedited Reporting to the Food and Drug Administration**

If the study is being conducted under an IND, the Sponsor-Investigator is responsible for determining whether or not the suspected adverse reaction meets the criteria for expedited reporting in accordance with Federal Regulations (21 CFR §312.32).

The Investigator must report in an IND safety report any suspected adverse reaction that is both serious and unexpected. The Sponsor-Investigator needs to ensure that the event meets all three definitions:

- Suspected adverse reaction (as defined in 6.1.30)
- Unexpected (as defined in 0)
- Serious (as defined in 6.1.5)

If the adverse event does not meet all three of the definitions, it should not be submitted as an expedited IND safety report.

The timeline for submitting an IND safety report to FDA is no later than **15 calendar days** after the Investigator determines that the suspected adverse reaction qualifies for reporting (21 CFR 312.32(c)(1)).

Any unexpected fatal or life-threatening suspected adverse reaction will be reported to FDA no later than **7 calendar days** after the Investigator's initial receipt of the information (21 CFR 312.32(c)(2)).

Any relevant additional information that pertains to a previously submitted IND safety report will be submitted to FDA as a Follow-up IND Safety Report without delay, as soon as the information is available (21 CFR 312.32(d)(2)).

#### 8 Statistical Considerations and Evaluation of Results

## 8.1 Study Endpoints

Primary endpoints:

- PSMA PET results for regional nodal disease.
- Nodal histology results from prostatectomy.

#### 8.1.1 Randomization

There will be no randomization performed. There will be no blinding performed.

## 8.2 Determination of Sample Size and Accrual Rate

#### 8.2.1 Sample Size and Power Estimate

Across all sites, the estimated sample size will be 271 patients in total to adequately power the primary aim. Our power analysis will be based on the comparison of sensitivity between conventional imaging and PSMA PET. With a power of 80% and a significance level of 0.01, we will require a sample size of 61 patients with nodal metastases. Given the assumptions below we will need to enroll a total of 271, although only those undergoing prostatectomy will be included for analysis (203 patients).

- i) 30% of intermediate to high-risk patients have nodal metastases at prostatectomy.
- ii) 25% of patients will not undergo the planned prostatectomy. Patients that do not undergo prostatectomy will not be included in the analysis population, and will not undergo central imaging review.
- iii) Conventional imaging has a 45% detection sensitivity for nodal metastases on a per patient basis (2).
- iv) PSMA PET has a 65% detection sensitivity for nodal metastases on a per patient basis.

#### 8.2.2 Accrual estimates

At all sites, we anticipate enrolling 300 patients in total. 300 patients will be enrolled at UCSF.

#### 8.3 Analyses Plans

## 8.3.1 Analysis Population

All patients that undergo prostatectomy and have histology correlates will be included in the analysis for the primary endpoint.

## 8.3.2 Analysis of Primary Endpoint

a) Imaging interpretation <sup>68</sup>Ga-PSMA-11 PET:

PET images will initially be interpreted by a board certified nuclear medicine physician or a board certified radiologist experienced in reading PET at the time of the imaging study at the institution that the study is being performed. These interpretations will not be used for final evaluation. Imaging data will be anonymized and collected at a central site. PET data will be interpreted by three different readers in a random order at separate reading sessions. Cross sectional imaging from the PET will be available for anatomic correlate. Final reads for each patient will be interpreted as positive or negative for the presence of pelvic nodal disease, and positive or negative for the presence of osseous metastatic disease and soft tissue metastases outside of the pelvis. <sup>68</sup>Ga-PSMA PET reading training set and guides will be provided and completion of this training will be required for all central review readers.

Visual interpretation of PET data:

Regions of suspected disease will be graded on a two-point scale by each reader (0=Negative or 1=Positive). A region will be judged as positive if at least one lesion in this region is visually positive.

- i) Lymph nodes will be considered positive if the <sup>68</sup>Ga-PSMA-11 uptake is focal and greater than adjacent background. Pelvic lymph nodes will be subclassified according to their localization as follows: R/L obturator, R/L external iliac, R/L internal iliac and other (total of 7 subgroups).
- ii) Visceral lesions will be considered positive if the <sup>68</sup>Ga-PSMA-11 uptake is focal and greater than physiologic background activity of the involvement organ or anatomic site.
- iii) Bone lesions will be considered positive if the <sup>68</sup>Ga-PSMA-11 uptake is focal and greater than physiologic bone marrow.
- b) Pathology analysis: Specimens from prostatectomy will be evaluated for the presence of nodal metastasis. This will be reported on a per patient basis as positive or negative.
  - i) Nodes will be marked by location per site specific protocol. For example if the urologist removed left and right nodal regions separately, then that patient will have two nodal regions (left/right). If a different surgeon removes nodes in six groups (bilateral internal/external/obturator nodes), then that patient will have six nodal regions that will be analyzed.

- ii) Although not routinely performed during standard practice, immunohistochemical staining for PSMA of tumor specimens (primary and lymph node metastases) may be performed, but is not required for this study.
- iii) The number of nodes counted on pathology will also be recorded.
- c) Analysis plan for Primary Aim 1: For this study to reach success, two out of the three readers will have to demonstrate a detection sensitivity of 65% or greater for nodal metastases. Additionally, two out of the three readers will have to demonstrate a detection specificity of 90% or greater for regional nodal metastases based upon region as defined below on a per patient level. The sensitivity, specificity, positive and negative predictive value of PSMA-11 PET for the detection on a per patient basis will be determined using the below criteria:
  - i) True positive patient:
    - (1) PSMA-11 PET positive for regional nodes; pathology at prostatectomy positive for regional nodes. Region will be defined by the granularity used by the urologist at time of prostatectomy. Sensitivity will be calculated at a patient level by region, meaning that one correct region would make a true positive on a patient level. Only one node needs to correspond between imaging and pathology for a patient to be considered a true positive.
    - (2) PSMA-11 PET positive for regional nodes, pathology negative for regional nodes, imaging after prostatectomy demonstrates node was not removed at surgery, and follow-up biopsy or imaging demonstrates presence of nodal disease.
      - (a) Criteria for positive node on follow-up imaging: imaging within 3-12 months, the node decreases by more than 30% (for patients undergoing systemic treatment or focal therapy at this site) or increase by more than 20% in short axis diameter in the absence of treatment (with a minimum of 3 mm in change in size).
  - ii) True negative patient:
    - (1) PSMA-11 PET negative for regional nodes; pathology at prostatectomy negative for regional nodes.
  - iii) False positive patient:
    - PSMA-11 PET positive for regional nodes, pathology at prostatectomy is negative, and imaging after prostatectomy demonstrates that node is no longer present.
    - (2) PSMA-11 PET positive for regional node, but pathology at prostatectomy is positive for node but in a different nodal region than that node seen on PSMA PET.
  - iv) False negative patient:
    - (1) PSMA-11 PET negative for regional nodes, but pathology at prostatectomy is positive.
  - v) Non-evaluable:

- (1) PSMA-11 PET positive for regional nodes, pathology negative for regional nodes, imaging after prostatectomy demonstrates node was not removed at surgery, and no definitive follow-up is available.
- (2) Patients with extrapelvic nodal metastases will not be included in this analysis if patients do not undergo prostatectomy.

## 8.3.3 Analysis of Secondary Endpoints

- a) Analysis plan for Secondary Endpoint 1: We will report the sensitivity, specificity, positive and negative predictive value of PSMA PET over all imaged regions as well as broken down by the following regions: extra-pelvic nodal metastases, visceral metastases and osseous metastases. Follow-up for extra-pelvic nodal metastases, visceral metastases and osseous metastases are defined as below:
  - i) <u>Lymph nodes</u> will be assessed by change in size. <sup>68</sup>Ga-PSMA-11 positive lymph nodes will be considered:
    - (1) True positive:
      - If on follow-up imaging within 3-12 months, lymph nodes seen on CT or MRI decrease by more than 30% (for patients undergoing systemic treatment of focal therapy at this site) or increase by more than 20% in short axis diameter (with a minimum of 3 mm in change in size).
      - If patients with solitary lymph node regions show a decrease of PSA by greater than 50% after targeted treatment (i.e. external beam radiation) and the lymph nodes do not change in size (less than 30% decrease or less than 20% increase in short axis diameter).
    - (2) False positive:
      - If on follow-up imaging within 3-12 months, sites of initial<sup>68</sup>Ga-PSMA-11 positive lymph node lesions seen on CT or MRI decrease by more than 30% without systemic therapy or focal therapy at this site.
      - If <sup>68</sup>Ga-PSMA-11 positive lymph node lesions do not meet the criteria for above false positive or true positive findings.
  - ii) <u>Visceral lesions (non-lymph node soft tissue or organ)</u> will be assessed by change in size. 68Ga-PSMA-11 positive visceral lesions will be considered:
    - (1) True positive:
      - If on follow-up imaging within 3-12 months, visceral lesions seen on CT or MRI decrease by 30% (for patients undergoing systemic treatment of focal therapy at this site) or increase by 20% in largest diameter.
      - If patients with solitary visceral metastasis show a decrease of PSA by greater than 50% after targeted treatment (i.e. external beam radiation) and lesions do not change in size (less than 30% decrease or 20% increase in largest diameter).
    - (2) False positive:

- If on follow-up imaging within 3-12 months, sites of initial<sup>68</sup>Ga-PSMA-11 positive visceral lesions seen on CT or MRI decrease by more than 30% without systemic therapy or focal therapy at this site.
- If <sup>68</sup>Ga-PSMA-11 positive visceral lesions do not meet the criteria for above false positive or true positive findings.
- iii) <sup>68</sup>Ga-PSMA-11 positive bone lesions will be considered:
  - (1) True positive:
    - If there was a corresponding positive sclerotic lesion on the CT portion of the <sup>68</sup>Ga-PSMA-11 PET in the same location as the PSMA uptake.
    - If there is focal uptake seen in the same location as the PSMA uptake on the baseline bone scan performed within one month of <sup>68</sup>Ga-PSMA-11 PET.
    - If there is a lesion noted in the same location as the PSMA uptake on the initial MRI performed within one month of <sup>68</sup>Ga-PSMA-11 PET.
    - If within 12 months follow-up CT demonstrates development of sclerosis in the same location as the PSMA uptake.
    - If within 12 months follow-up MRI demonstrates a new bone lesion in the same location as the PSMA uptake.
    - If within 12 months follow-up bone scan demonstrates new focal uptake in the same location as the PSMA uptake.
  - (2) False positive:
    - If <sup>68</sup>Ga-PSMA-11 positive bone lesions do not meet the criteria for true positive findings.
- iv) Histopathology correlation: for lesions that have biopsy correlation, we will use the following criteria to determine positive and negative lesions:
  - (1) <u>Positive HP/Biopsy</u>: Confirmed sites of metastatic or tumor involvement by histopathology/biopsy will be discussed with the responsible physician/surgeon.
  - (2) <u>Negative Biopsy</u>: Patients with suspected tumor recurrence on 68Ga-PSMA-11 PET with negative histopathology/biopsy will be handled as outlined below:
    - (a) Lymph nodes:
      - For patients undergoing nodal dissection: Patients will be rescanned with dedicated CT or MRI to determine if the suspicious <sup>68</sup>Ga-PSMA-11 positive node was removed.
        - If <sup>68</sup>Ga-PSMA-11 positive lymph node is still present, a repeat biopsy can be pursued if clinically feasible and applicable, or follow-up using imaging as described above will be performed.
        - If the corresponding node was removed, then this will be considered a False Positive.

- For patients undergoing needle biopsy: Images of the procedure will be reviewed to determine if the correct node was biopsied.
  - If the correct node was biopsied, then a negative biopsy will be considered a False Positive.
  - If the incorrect node was biopsied, then follow-up imaging as described above will be performed.
- (b) Bone lesions: Given the high rate of false negative biopsies for osseous metastases in patients with prostate cancer, patients with negative bone biopsies of PSMA PET positive lesions will be further evaluated:
  - If pathology demonstrates an alternative diagnoses that is known to be PSMA positive (eg Renal Cell Carcinoma metastases, Paget's disease), then this will be considered a False Positive.
  - If pathology is indeterminate, then follow-up imaging as described above will be performed to determine if the lesion is a True Positive or False Positive.
- (c) Additionally a repeat <sup>68</sup>Ga-PSMA-11 can also be obtained, as allowable, in addition to repeat conventional imaging (CT and/or MRI) in cases of negative biopsy to determine if the biopsy was true negative or false negative.
- b) Safety: Safety will be reported descriptively as rates of patient reported adverse events. Additionally, adverse events will be characterized and quantified by CTCAE 4.03.

## 8.3.4 Analysis of Exploratory Endpoints

PPVs on a per-patient and per-region-basis of <sup>68</sup>Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy and conventional imaging follow-up will be calculated and reported along with the corresponding two-sided 95% confidence intervals. The paired McNemar's test will be used to compare the PPVs of <sup>68</sup>Ga-PSMA-11 PET imaging to the PPVs of conventional imaging.

Sensitivity, specificity, and NPVs on a per-patient basis of <sup>68</sup>Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy will be summarized in tabular format. Furthermore, the positive and negative likelihood ratios (LR+ and LR-) will be calculated and reported. Ninety-five confidence intervals of sensitivity, specificity, and NPV will be calculated using the Wilson score method. The comparisons of sensitivity, specificity, and NPV on a per-patient basis of <sup>68</sup>Ga-PSMA-11 PET imaging will be compared to of sensitivity, specificity, and NPV on a per-patient basis of conventional imaging using a paired McNemar's test.

Detection rates on a per-patient basis of <sup>68</sup>Ga-PSMA-11 PET stratified by PSA value (0.2 - <0.5, 0.5 - <1.0, 1.0 - <2.0, 2.0 - <5.0, 5.0) will be summarized in tabular format and compared between PSA strata using chi-square analysis. The impact of <sup>68</sup>Ga-PSMA-11 PET on clinical management in BCR patients will be evaluated using descriptive statistics.

## 9 Study Management

## 9.1 Pre-study Documentation

This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki as stated in 21 CFR §312.120(c)(4); consistent with GCP and all applicable regulatory requirements.

Before initiating this trial, the Investigator will have written and dated approval from the Institutional Review Board for the protocol, written informed consent form, subject recruitment materials, and any other written information to be provided to subjects before any protocol related procedures are performed on any subjects.

The clinical investigation will not begin until either FDA has determined that the study under the Investigational Drug Application (IND) is allowed to proceed or the Investigator has received a letter from FDA stating that the study is exempt from IND requirements.

## 9.2 Institutional Review Board Approval

The protocol, the proposed informed consent form, and all forms of participant information related to the study (e.g. advertisements used to recruit participants) will be reviewed and approved by the UCSF CHR (UCSF Institutional Review Board). Prior to obtaining CHR approval, the protocol must be approved by the Helen Diller Family Comprehensive Cancer Center Site Committee and by the Protocol Review Committee (PRC). The initial protocol and all protocol amendments must be approved by the IRB prior to implementation.

#### 9.3 Informed Consent

All participants must be provided a consent form describing the study with sufficient information for each participant to make an informed decision regarding their participation. Participants must sign the CHR-approved informed consent form prior to participation in any study specific procedure. The participant must receive a copy of the signed and dated consent document. The original signed copy of the consent document must be retained in the medical record or research file.

## 9.4 Changes in the Protocol

Once the protocol has been approved by the UCSF CHR, any changes to the protocol must be documented in the form of an amendment. The amendment must be signed by the Investigator and approved by PRC and the CHR prior to implementation.

If it becomes necessary to alter the protocol to eliminate an immediate hazard to patients, an amendment may be implemented prior to CHR approval. In this circumstance, however, the Investigator must then notify the CHR in writing within five (5) working days after implementation. The Study Chair and the UCSF study team will be responsible for updating any participating sites.

## 10 Protection of Human Subjects

#### 10.1 Protection of Privacy

Patients will be informed of the extent to which their confidential health information generated from this study may be used for research purposes. Following this discussion, they will be asked to sign the HIPAA form and informed consent documents. The original signed document will

become part of the patient's medical records, and each patient will receive a copy of the signed document. The use and disclosure of protected health information will be limited to the individuals described in the informed consent document.

#### References

- 1. Edwards BK, Noone A-M, Mariotto AB, et al. Annual Report to the Nation on the status of cancer, 1975-2010, featuring prevalence of comorbidity and impact on survival among persons with lung, colorectal, breast, or prostate cancer. Cancer. 2014;120:1290–1314.
- 2. Oyen RH, Van Poppel HP, Ameye FE, Van de Voorde WA, Baert AL, Baert LV. Lymph node staging of localized prostatic carcinoma with CT and CT-guided fine-needle aspiration biopsy: prospective study of 285 patients. 1994;190:315–322.
- 3. Contractor K, Challapalli A, Barwick T, et al. Use of [11C]choline PET-CT as a noninvasive method for detecting pelvic lymph node status from prostate cancer and relationship with choline kinase expression. Clin Cancer Res. 2011;17:7673–7683.
- 4. Price DT, Coleman RE, Liao RP, Robertson CN, Polascik TJ, DeGrado TR. Comparison of [18 F]fluorocholine and [18 F]fluorodeoxyglucose for positron emission tomography of androgen dependent and androgen independent prostate cancer. J Urol. 2002;168:273—280.
- 5. Castellucci P, Ceci F, Graziani T, et al. Early biochemical relapse after radical prostatectomy: which prostate cancer patients may benefit from a restaging 11C-Choline PET/CT scan before salvage radiation therapy? J Nucl Med. 2014;55:1424–1429.
- 6. Brogsitter C, Zöphel K, Kotzerke J. 18F-Choline, 11C-choline and 11C-acetate PET/CT: comparative analysis for imaging prostate cancer patients. Eur J Nucl Med Mol Imaging. 2013;40 Suppl 1:S18–S27.
- 7. Picchio M, Spinapolice EG, Fallanca F, et al. [11C]Choline PET/CT detection of bone metastases in patients with PSA progression after primary treatment for prostate cancer: comparison with bone scintigraphy. Eur J Nucl Med Mol Imaging. 2011;39:13–26.
- 8. Souvatzoglou M, Krause BJ, Pürschel A, et al. Influence of (11)C-choline PET/CT on the treatment planning for salvage radiation therapy in patients with biochemical recurrence of prostate cancer. Radiother Oncol. 2011;99:193–200.
- 9. Castellucci P, Fuccio C, Rubello D, et al. Is there a role for <sup>11</sup>C-choline PET/CT in the early detection of metastatic disease in surgically treated prostate cancer patients with a mild PSA increase. Eur J Nucl Med Mol Imaging. 2011;38:55–63.
- 10. Giovacchini G, Picchio M, Scattoni V, et al. PSA doubling time for prediction of [(11)C]choline PET/CT findings in prostate cancer patients with biochemical failure after radical prostatectomy. Eur J Nucl Med Mol Imaging. 2010;37:1106–1116.
- 11. Fuccio C, Castellucci P, Schiavina R, et al. Role of 11C-choline PET/CT in the restaging of prostate cancer patients showing a single lesion on bone scintigraphy. Ann Nucl Med. 2010;24:485–492.
- 12. Seltzer MA, Barbaric Z, Belldegrun A, et al. Comparison of helical computerized tomography, positron emission tomography and monoclonal antibody scans for

- evaluation of lymph node metastases in patients with prostate specific antigen relapse after treatment for localized prostate cancer. J Urol. 2005;162:1322–1328.
- 13. Kahn D, Williams RD, Manyak MJ, et al. 111Indium-capromab pendetide in the evaluation of patients with residual or recurrent prostate cancer after radical prostatectomy. The ProstaScint Study Group. J Urol. 1998;159:2041–6–discussion2046–7.
- 14. Manyak MJ, Hinkle GH, Olsen JO, et al. Immunoscintigraphy with indium-111-capromab pendetide: evaluation before definitive therapy in patients with prostate cancer. Urology. 1999:54:1058–1063.
- 15. Raj GV, Partin AW, Polascik TJ. Clinical utility of indium 111-capromab pendetide immunoscintigraphy in the detection of early, recurrent prostate carcinoma after radical prostatectomy. Cancer. 2002;94:987–996.
- 16. Aparici CM, Carlson D, Nguyen N, Hawkins RA, Seo Y. Combined SPECT and Multidetector CT for Prostate Cancer Evaluations. Am J Nucl Med Mol Imaging. 2012;2:48–54.
- 17. Afshar-Oromieh A, Zechmann CM, Malcher A, et al. Comparison of PET imaging with a (68)Ga-labelled PSMA ligand and (18)F-choline-based PET/CT for the diagnosis of recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2014;41:11–20.
- 18. Afshar-Oromieh A, Avtzi E, Giesel FL, et al. The diagnostic value of PET/CT imaging with the (68)Ga-labelled PSMA ligand HBED-CC in the diagnosis of recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2015;42:197–209.
- 19. Eiber M, Maurer T, Souvatzoglou M, et al. Evaluation of Hybrid <sup>68</sup>Ga-PSMA Ligand PET/CT in 248 Patients with Biochemical Recurrence After Radical Prostatectomy. J Nucl Med. Society of Nuclear Medicine. 2015;56:668–674.
- 20. Ceci F, Uprimny C, Nilica B, et al. (68)Ga-PSMA PET/CT for restaging recurrent prostate cancer: which factors are associated with PET/CT detection rate? Eur J Nucl Med Mol Imaging. 2015;42:1284–1294.
- 21. van Leeuwen PJ, Stricker P, Hruby G, et al. (68) Ga-PSMA has a high detection rate of prostate cancer recurrence outside the prostatic fossa in patients being considered for salvage radiation treatment. BJU Int. 2016;117:732–739.

Version date: 2018.06.08

Protocol CC#: 16559



# **Appendices**

# Appendix 1 Performance Status Criteria

| ECOG Performance Status Scale | | Karnofsky Performance Scale | |
|---|---|---|---|
| Grade | Descriptions | Percent | Description |
| Normal activity Fully active, able to carry on all | | 100 | Normal, no complaints, no evidence of disease |
| | pre-disease performance without restriction | 90 | Able to carry on normal activity; minor signs or symptoms of disease |
| 1 | Symptoms, but ambulatory Restricted in physically strenuous activity, but ambulatory and able | 80 | Normal activity with effort; some signs or symptoms of disease |
| | to carry out work of a light or sedentary nature (e.g., light housework, office work) | | Cares for self, unable to carry on normal activity or to do active work |
| 2 | 2 In bed < 50% of the time Ambulatory and capable of all self-care, but unable to carry out any work activities Up and about more than 50% of waking hours | | Requires occasional assistance, but is able to care for most of his/her needs |
| | | | Requires considerable assistance and frequent medical care |
| 3 | In bed > 50% of the time | 40 | Disabled, requires special care and assistance |
| | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours | | Severely disabled, hospitalization indicated Death not imminent |
| 4 | 100% bedridden | 20 | Very sick, hospitalization indicated |
| | Completely disabled | | Death not imminent |
| Cannot carry on any self-care Totally confined to bed or chair | | 10 | Moribund, fatal processes progressing rapidly |
| 5 | Dead | 0 | Dead |

# Appendix 2 Schedule of procedures

| Table 1.1 Schedule of Study Procedures and Assessments | | | |
|---|---|---|---|
| Period/<br>Procedure | Screening | Imaging day 1 | One day post imaging |
| Study Day/Visit Day | -30 to 1 | 1 | 2-4 |
| Informed consent | Х | | |
| Laboratory values, history from medical record | Х | | |
| Pre-survey | X | | |
| Performance status | X | | |
| Blood Pressure, HR | Х | Х | |
| Imaging Procedure | | | |
| Ga-68 PSMA-11 | | Х | |
| PET/CT or PET/MRI | | Х | |
| Follow-up | | | |
| Adverse event reporting | | | X |

## **Appendix 3 (flow chart)**

